CLINICAL TRIAL: NCT03701152
Title: Comparison Between Two Different Protocols of Negative Pressure Therapy for Healing of Chronic Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Ashraf Hassan, Professor, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001669
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Ulcers; Negative Pressure Therapy
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure therapy (Experimental): Negative pressure therapy topical application using negative pressure therapy sub atmospheric pressure Continuous course
  Interventions: Device: Negative pressure therapy
- Investigator (Experimental): Negative pressure therapy topical application using negative pressure therapy sub atmospheric pressure Splitted course
  Interventions: Device: Negative pressure therapy

INTERVENTIONS:
Device: Negative pressure therapy — Negative pressure therapy at sub atmospheric level

SUMMARY:
Negative Pressure Wound Therapy (NPWT), is a non invasive wound management tool which develops from negative pressure being applied to the wound. This promotes healing through the removal of infectious materials and enhancing granulation tissue formation. NPWT eases debridement as well as promoting healing of different types of wounds.

DETAILED DESCRIPTION:
Assessment of wound surface area was done by a graded plastic sheet and a metric graph paper, by counting the complete squares of the metric graph paper, while the wound size was done by using a 10 cm syringe filled with dermazin cream and filling the wound with it.

Negative pressure device: VAC system 125mmhg (KCI negative pressure equipment).

Wound surface area tracing tools:

* Sterilized transparent film.
* Fine tipped transparent marker.
* Carbon and a white A4 papers.
* Metric graph paper (1mm²).

Wound volume assessment procedure:

* Using a syringe of ten cubic centimeters filled with dermazin cream.
* The wound is filled with the cream
* The amount of cream injected into the wound was detected in cubic centimeters.

ELIGIBILITY:
Inclusion Criteria:

* They were free from immune deficiency diseases or collagen diseases.
* All patients were homeostasis.
* All patients were medically stable.
* All cases were chronic and did not heal with other treatment methods

Exclusion Criteria:

* 1. Malignancies or receiving radiotherapy. 2. Dermatological diseases. 3. Deep venous thrombosis. 4. Renal failure. 5. Immunosuppressant or anticonvulsants therapies.

Ages: 27 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Wound surface area | 8 weeks
Wound size | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, Egypt

REFERENCES:
- [Derived] Mohammed AH, Hamed SA, Abdelghany AI. Comparison between two different protocols of negative pressure therapy for healing of chronic ulcers. J Tissue Viability. 2020 Feb;29(1):37-41. doi: 10.1016/j.jtv.2019.10.003. Epub 2019 Oct 25. PMID 31677995